CLINICAL TRIAL: NCT07323056
Title: Sacituzumab Tirumotecan and Limertinib for Conversion Therapy in Locally Advanced Potentially Resectable EGFR-mutant Non-small Cell Lung Cancer: A Prospective, Single-arm, Exploratory Clinical Study
Brief Title: Neoadjuvant Sacituzumab Tirumotecan and Limertinib for Potentially Resectable Stage Ⅲ EGFR-mutant Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-037
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: EGFR-mutant Non-small Cell Lung Cancer; Potentially Resectable
Keywords: non-small cell lung cancer; EGFR-mutant; Sacituzumab Tirumotecan; Limertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical treatment after targeted therapy combined with chemotherapy (Experimental)
  Interventions: Drug: Sacituzumab Tirumotecan and Limertinib

INTERVENTIONS:
Drug: Sacituzumab Tirumotecan and Limertinib — Sacituzumab Tirumotecan injection is administered once every two weeks for a total of six treatments. Sacituzumab Tirumotecan injection: 4 mg/kg, intravenous infusion, Q2W. Limertinib is administered for 12 weeks. Limertinib: standard dose, oral, Qd. After the completion of the neoadjuvant treatment cycle, enhanced chest CT and other evaluations are conducted. The feasibility of radical surgery is assessed by MDT. Patients who are eligible for surgery will undergo surgical treatment, and the treatment plan for those who are not eligible for surgery will be determined after discussion by MDT.

SUMMARY:
This study is a prospective, single-arm, exploratory clinical research aimed at evaluating the efficacy and safety of lucetamab in combination with leucovorin in the conversion therapy of locally advanced potentially resectable EGFR mutation-positive non-small cell lung cancer, providing more robust clinical evidence for the improvement of treatment modalities for EGFR-mutated locally advanced NSCLC. At the same time, it seeks to identify biomarkers that can predict the therapeutic effect of the combination of lucetamab and leucovorin, offering more precise guidance for the selection of clinical treatment plans and enabling patients to receive the optimal treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form
* The age of the subjects is over 18 years old
* Patients with non-small cell lung cancer (NSCLC) with EGFR mutation confirmed by pathology
* Confirmed as locally advanced NSCLC (IIIA, IIIB, IIIC) by chest CT, PET-CT or/and EBUS, and MDT discussion concludes that immediate local surgery is not suitable
* Have not received systematic anti-tumor treatment before
* The researcher confirms at least one measurable lesion according to RECIST 1.1 criteria
* Good lung function and able to tolerate surgical treatment
* ECOG score is 0 to 1

Exclusion Criteria:

* Allergy to Sacituzumab Tirumotecan or any of its excipients
* Patients allergic to Limertinib or any of its excipients
* Patients with a history of other primary tumors; patients with a history of allogeneic organ transplantation
* Major surgery within 4 weeks before the first dose (excluding diagnostic biopsy)
* Patients with drug addiction such as drug abuse, long-term alcohol abuse, AIDS or HIV carriers
* Patients with active or previously had and may recur autoimmune diseases
* Currently receiving systemic hormone therapy (such as equivalent to more than 10 mg of prednisone per day or any other form of immunosuppressive therapy within 14 days before the first dose)
* Patients who have received any EGFR-TKI or TROP2 ADC treatment before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Perioperative

SECONDARY OUTCOMES:
Major pathologic response (MPR) rate | Perioperative
Objective response rate (ORR) | Up to 3 months
Event-free suvival (EFS) | Up to 60 months
Overall suvival (OS) | Up to 60 months
R0 resection rate | Perioperative
Incidence of treatment discontinuation due to AE/SAE | Up to 3 months
Treatment-related adverse event (TRAE) | Up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether IPD is available to other researchers only after the paper is published.